CLINICAL TRIAL: NCT03106844
Title: The ICON Study: Inflammatory Bowel Disease and Recurrent Clostridium Difficile Infection: Outcomes After Fecal Microbiota Transplantation
Brief Title: The ICON Study: Outcomes After FMT for Patients With IBD and CDI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Indiana University (Other); Icahn School of Medicine at Mount Sinai (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ravikoff Allegretti, Principle Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000386
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Bowel Diseases; Clostridium Difficile Infection
Keywords: FMT; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients in this study will receive Fecal Microbiota Tranplantation
  Interventions: Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Patients with at least 2 episodes of CDI and IBD will undergo a single FMT
  Other Names: FMT

SUMMARY:
In this study the investigators will evaluate patients with IBD and and at least 2 confirmed c.difficile infections who will be undergoing FMT. The investigators will assess patients before FMT and then follow patients prospectively post FMT at week 1, 8 and 12 to assess for recurrence of c.difficile infection and IBD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater
* Confirmed recurrent CDI by positive PCR or EIA toxin test defined at ≥ 2 episodes and vancomycin failure within one year with the most recent being within the past 3 months.
* Confirmed diagnosis of IBD with colonic involvement (ulcerative colitis, Crohn's colitis or ileocolitis or indeterminate colitis) for ≥ 3 months
* Undergoing FMT via colonoscopy for CDI as part of standard medical care

Exclusion Criteria:

* Unable or unwilling to undergo a colonoscopy
* Inpatient status
* Anticipated immediate or upcoming surgery within 30 days
* Need for continued non-anti-CDI antibiotic therapy
* History of total or subtotal proctocolectomy
* Isolated ileal or small bowel disease
* Pregnancy or lactation
* Female patients who are pregnant or breastfeeding or plan to become pregnant in the next 6 months.
* Patients who are unable to give informed consent
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Severe food allergy (anaphylaxis or anaphylactoid-like reaction)
* Life expectancy < 6 months
* Unable to adhere to protocol requirements
* Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines that it will put the subject at greater risk from FMT
* Known concurrent HIV, Hepatitis B or C infection
* Concurrent PSC
* Patients with WBC< 3.0 x109th/L at baseline
* Patients with platelet count < 100 x109th/L
* Patients with initial elevation of AST or ALT > 1.5 times above normal limit at baseline
* Non - steroidal anti-inflammatory medications (NSAIDs) as long-term treatment, defined as use for at least 4 days a week each month
* Treatment with vancomycin or metronidazole for more then 60 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Allegretti, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 43 [21 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Calprotectin [Mean (Standard Deviation); unit: mg/L] | 5.3 (8.7)
Baseline C-Reactive Protein [Mean (Standard Deviation); unit: ug/g] | 1919.6 (2432.3)
Average Bowel Movements [Mean (Standard Deviation); unit: bowel movements] | 5.2 (4.0)
Average Bristol Score [Mean (Standard Deviation); unit: units on a scale] — Range 1-7. Low scores represent hard stools and high numbers represent liquid stools
  units on a scale | 5.6 (1.1)
Average Complete Mayo [Mean (Standard Deviation); unit: units on a scale] — Range 0-12. The score is a ulcerative colitis disease activity assessement and has 4 components: bowel movements, rectal bleeding, physical global assessment and endoscopy score. Each component ranges from 0-3. The scores from each subsection are added together to get the total score. Low scores indicate inactive disease. High scores indicate active disease.
  units on a scale | 5.6 (3.3)
Average Partial Mayo [Mean (Standard Deviation); unit: units on a scale] — Range 0-9. The score is a ulcerative colitis disease activity assessment and has 3 components: bowel movements, rectal bleeding, and physical global assessment. Each component ranges from 0-3. The scores from each subsection are added together to get the total score. Low scores indicate inactive disease. High scores indicate active disease.
  units on a scale | 4.2 (2.1)
Average Harvey Bradshaw Index [Mean (Standard Deviation); unit: units on a scale] — This is a disease activity index for Crohn's disease. Components include: general well being [score 0-4] abdominal pain [score 0-3], number of liquid stools, abdominal mass [score 0-3], and complications of disease [score 0-8]. The score if each component is added together to get the total score [Range 0 to 18] The upper range is open ended as the number of liquid stools will vary by patient. HBI < 5 is defined as clinical remission, HBI between 5 and 7 as mild disease, HBI between 8 and 16 as moderate disease, and HBI > 16 as severe disease.
  units on a scale | 5.8 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With FMT Failure
Description: Recurrence of c.diffile infection
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 49
Participants | 4

2. Secondary Outcome: Participants Colonized With C.Difficile
Description: asymptomatic patients with positive stool testing for c.difficile via polymerase chain reaction testing
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 49
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through week 26 (6 months)
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=50)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Subject required blood transfusion due to severe anemia. This AE was determined unrelated to treatment and due to previous condition.
IBD Flare (Gastrointestinal disorders) | 1 (1) — The subject had IBD flare that required hospitalization. This was deemed to be unrelated to study treatment and reported at the week 8 follow-up.
IBD Flare (Gastrointestinal disorders) | 1 (1) — Patient was experiencing Diarrhea and a fever due to an IBD flare. Subject was admitted to hospital and treated with an IV of omnipaque and later discharged.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=50)
Diarrhea (Gastrointestinal disorders) | 22
Rectal Bleeding (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Fever (General disorders) | 5
Fatigue (General disorders) | 3
Heart Burn (Gastrointestinal disorders) | 2
Chills (General disorders) | 2
Migraine (Nervous system disorders) | 2
Yeast Infection (Renal and urinary disorders) | 2
Constiption (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03106844/Prot_SAP_000.pdf